CLINICAL TRIAL: NCT05108584
Title: The Intubation Procedure in COVID-19 Pandemic
Brief Title: Intubation in Coronavirus Disease 19 With Level 3 PPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, MD, PhD, Anesthesiologist Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IndonesiaU120
Record Dates: First submitted 2021-10-18; First posted 2021-11-05 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Intubation Complication
Keywords: COVID-19; Intubation process; Personal protective equipment (PPE); Laryngoscope
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 - Level 3 PPE and video laryngoscope (Experimental): Pre-anesthesia visit aims to assess the participant's physical status based on the American Society of Anesthesiologists score and assessment of the airway. Researcher then explained about the study and plan for anesthesia using an endotracheal tube and personal protective equipment according to the group. While in the operating room, the intubation operator was assisted by an assistant who already used appropriate PPE. Coveralls or hazmat suits and surgical gowns used must match the size. The intubation operator was resident of Anesthesiology and Intensive Therapy study program (stage II) and accompanied by an independent resident (stage III) and an anesthesiologist on duty. The operator used level 3 PPE (coverall jumpsuit, face shield, goggles, N95 mask, surgical mask, boot, scrub, and two layered gloves) and video laryngoscope for intubation of the participants. Researcher was in charge for recording time and event during the intubation process according to the study form.
  Interventions: Procedure: PPE Level 3 and Video Laryngoscope
- Group 2 - Level 3 PPE and direct laryngoscope (Experimental): Pre-anesthesia visit aims to assess the participant's physical status based on the American Society of Anesthesiologists score and assessment of the airway. Researcher then explained about the study and plan for anesthesia using an endotracheal tube and personal protective equipment according to the group. While in the operating room, the intubation operator was assisted by an assistant who already used appropriate PPE. Coveralls or hazmat suits and surgical gowns used must match the size. The intubation operator was resident of Anesthesiology and Intensive Therapy study program (stage II) and accompanied by an independent resident (stage III) and an anesthesiologist on duty. The operator used level 3 PPE (coverall jumpsuit, face shield, goggles, N95 mask, surgical mask, boot, scrub, and two layered gloves) and direct laryngoscope for intubation of the participants. Researcher was in charge for recording time and event during the intubation process according to the study form.
  Interventions: Procedure: PPE Level 3 and Direct Laryngoscope
- Group 3 - Level 2 PPE and direct laryngoscope (Experimental): Pre-anesthesia visit aims to assess the participant's physical status based on the American Society of Anesthesiologists score and assessment of the airway. Researcher then explained about the study and plan for anesthesia using an endotracheal tube and personal protective equipment according to the group. While in the operating room, the intubation operator was assisted by an assistant who already used appropriate PPE. Coveralls or hazmat suits and surgical gowns used must match the size. The intubation operator was resident of Anesthesiology and Intensive Therapy study program (stage II) and accompanied by an independent resident (stage III) and an anesthesiologist on duty. The operator used level 2 PPE (surgical gown/apron, face shield, goggles, N95 mask, surgical mask, boot, scrub, and two layered gloves) and video laryngoscope for intubation of the participants. Researcher was in charge for recording time and event during the intubation process according to the study form.
  Interventions: Procedure: PPE Level 2 and Direct Laryngoscope

INTERVENTIONS:
Procedure: PPE Level 3 and Video Laryngoscope — The operator used level 3 PPE and video laryngoscope for the intubation process
  Arms: Group 1 - Level 3 PPE and video laryngoscope
Procedure: PPE Level 3 and Direct Laryngoscope — The operator used level 3 PPE and direct laryngoscope for the intubation process
  Arms: Group 2 - Level 3 PPE and direct laryngoscope
Procedure: PPE Level 2 and Direct Laryngoscope — The operator used level 2 PPE and direct laryngoscope for the intubation process
  Arms: Group 3 - Level 2 PPE and direct laryngoscope

SUMMARY:
The World Health Organization (WHO) declared COVID-19 as a pandemic in April 2020. COVID-19 first discovered in Wuhan, China in December 2019. As of May 4th, 2020, the total number of patients in China was 82,880, the number of deaths was 4,633, the death rate was 3.7%. In Indonesia, until May 4th 2020, there were 11,192 confirmed cases of COVID-19 with a total of 845 deaths. High transmission and death due to the severe acute respiratory syndrome coronavirus 2, patients with respiratory failure symptoms were suspected of having COVID-19 until declared negative. A potential and continuing threatening complication is acute respiratory failure. Patient with Acute Respiratory Distress Syndrome (ARDS) require both respiratory support and oxygen therapy. The choosing of endotracheal intubation is generally indicated in moderate to severe ARDS. Apart from respiratory failure, endotracheal intubation is also commonly performed in patients undergoing surgical procedures under general anesthesia for the management of the patient's airway. To prevent transmission to medical personnel, intubation is carried out using PPE according to the guidelines. Guidance for intubation in COVID-19 patients is recommended to use a video laryngoscope because it offers several advantages such as assisting glottis visualization and making the intubation operator more distant from the patient's mouth when compared to direct laryngoscopes. This study aims to see the effect of using PPE and the type of laryngoscope on the intubation process carried out in the COVID-19 pandemic. This study is a preliminary study aimed at seeing the effect size of the recommended PPE use on the process and success of intubation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 59 years old
* Undergo elective or emergency surgery using general anesthesia with endotracheal tube
* BMI below 30 kg/m2

Exclusion Criteria:

* Airway difficulty as assessed by preoperative assessment
* Critical patients with unstable hemodynamics
* Suspected or confirmed COVID-19 with ASA 3-5

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Total duration of the intubation process | During the procedure
  The sum amount of time needed to complete an intubation process that includes preoxygenation duration, neuromuscular blocker action, laryngoscopy duration, and endotracheal tube position confirmation with ultrasound
Success of intubation process as assessed by number of trials | During the procedure
  The sum amount of trials needed to successfully place an endotracheal tube to the respiratory system
Safety as assessed by number of participants experiencing complications | During the procedure
  Number of participants who experience desaturation of oxygen (below 95%), airway injury, increased blood pressure (over 120/80 mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Dita Aditianingsih, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes